CLINICAL TRIAL: NCT05575778
Title: The Clinical Value of Quantitative Analysis of Peri-operative Foot Supply Through CT Perfusion in Patients With Critical Limb Ischemia
Brief Title: Peri-operative Foot CT Perfusion in CLI Patients
Acronym: POP-CLI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: 2022KW
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: computed tomographic perfusion — The recruited patients would complete both pre- and post-operative computed tomographic perfusion

SUMMARY:
To investigate the clinical value of quantitative analysis of peri-operative foot supply through CT perfusion in patients with critical limb ischemia

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old;
* CLI patients with Fontaine grade III-IV or Rutherford grade 4-6 and underwent a successful revascularization;
* Patients completed both pre- and post-operative CTP workups;
* Patients signed the informed consent form and be able to complete the clinical follow-up for 12 months.

Exclusion Criteria:

* Patients has participated in other clinical studies;
* Patients with Heart failure (NYHA III/IV)/right to left shunt heart disease/severe aortic and mitral insufficiency/acute coronary syndrome/malignant arrhythmia/severe pulmonary hypertension (pulmonary artery pressure at least 90 mmHg)/moderate to severe renal insufficiency (creatinine clearance rate<60 ml/min)
* Any allergic constitution;
* Pregnancy and childbirth;
* Life expectancy<12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with critical limb ischemia, who completed both pre- and post-operative CTP workups
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pre-operative computed tomographic perfusion parameters | 18months
  Pre-operative computed tomographic perfusion parameters, including peak intensity, time to peak, and etc, which would be obtained three days before revascularization.
Post-operative computed tomographic perfusion parameters | 18months
  Post-operative computed tomographic perfusion parameters, including peak intensity, time to peak, and etc, which would be obtained three days ater revascularization.
Alteration of computed tomographic perfusion parameters | 18months
  Alteration between post- (three days ater revascularization) and pre-operative (three days before revascularization) computed tomographic perfusion parameters

SECONDARY OUTCOMES:
Major adverse limb events | 12months
  Major adverse limb events included major amputation or acute limb ishchemia for vasular causes.
Major adverse cardiovascular events | 12months
  Major adverse cardiovascular events included myocardial infarction, ischemic stroke, or death from cadiovascular causes.

OTHER OUTCOMES:
All-cause deah | 12months
  All-cause deah during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Wan Zhang, PH.D., Principal Investigator — Huadong Hospital affiliated to Fudan University, Shanghai, China, 200040
Locations (1):
- Hua Dong Hospital Affiliated to Fu Dan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No